CLINICAL TRIAL: NCT06877117
Title: Exploring Nudging Strategies to Encourage Rectangular Collimation in Pediatric Dental Practice
Brief Title: Rectangular Collimation in Pediatric Dentistry
Acronym: RCPD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Varsha Lal, Principle Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 47738
Record Dates: First submitted 2025-03-04; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Behaviour Change; Nudging; Rectangular Colllimation in Pediatric Dentistry
MeSH Terms: interventions — Memory and Learning Tests

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Control Arm receives only didactic information and no nudges
- Pictorial Framing (Experimental): Written information is supplemented with pictorial nudges.
  Interventions: Behavioral: Pictorial Framing
- Traffic Light Color Coding (Experimental): Written information is supplemented with traffic light colour coding nudges.
  Interventions: Behavioral: Traffic Light Color Coding Framing

INTERVENTIONS:
Behavioral: Pictorial Framing — Visual aids illustrating collimation benefits
  Other Names: Behavioural; Prompt; Pictorial Nudging; Framing
  Arms: Pictorial Framing
Behavioral: Traffic Light Color Coding Framing — Decision cues using color-based risk indicators
  Other Names: Nudges; Framing; behavioral; prompt
  Arms: Traffic Light Color Coding

SUMMARY:
This project aims to investigate whether simple behavioural interventions, such as pictorial framing and traffic-light-color-coding, can positively influence pediatric dentists' decision-making in adopting rectangular collimation over round collimation for dental radiographs taken in clinical practice.

DETAILED DESCRIPTION:
1. Introduction Dental radiographs are essential in diagnosing oral conditions in pediatric patients. Despite the availability of rectangular collimation as a recommended radiation safety measure, many pediatric dentists continue to use round collimation, which results in unnecessary radiation exposure. This study explores whether nudging strategies-such as pictorial framing and traffic-light color coding-can influence pediatric dentists' decision-making to encourage the adoption of rectangular collimation.
2. Research Objectives

   This study aims to:

   Educate pediatric dentists on the benefits of rectangular collimation over round collimation.

   Assess current collimation practices among pediatric dentists. Evaluate whether behavioral nudging strategies influence pediatric dentists' willingness to adopt rectangular collimation.
3. Study Hypothesis Null Hypothesis: Nudging strategies (pictorial framing and traffic-light color coding) have no impact on pediatric dentists' willingness to adopt rectangular collimation.

   Alternative Hypothesis: The implementation of nudging strategies positively influences pediatric dentists to use rectangular collimation.
4. Methodology Study Design

   * A randomized, quantitative survey distributed online.
   * Three study groups:

1. Control Group (No nudging intervention) 2. Pictorial Framing Group (Visual aids illustrating collimation benefits) 3. Traffic-Light Color Coding Group (Decision cues using color-based risk indicators)

Participants Target Population: Pediatric dentists who are active members of the American Academy of Pediatric Dentistry (AAPD) in the U.S. and Canada.

Sample Size: As a one of its kind research project, the minimum for comparison is 30 participants in each sample group.

Data Collection A self-administered online survey conducted via REDCap. Survey distribution follows randomization of participants into the three groups.

Three e-mail invitations sent at two-week intervals over a six-week period.

Outcome Measures Primary Outcome: Change in willingness to adopt rectangular collimation. Secondary Outcome: Differences in responses across study groups.

Statistical Analysis Descriptive and comparative statistics using SPSS. Statistical significance set at p < 0.05.

5. Ethical Considerations Study approved by the University of Toronto Health Sciences Research Ethics Board.

Participants' responses are anonymous, and data security measures are in place.

6. Expected Impact This study will provide valuable insights into behavioral interventions for pediatric dentistry. If effective, nudging strategies could be incorporated into clinical guidelines to enhance radiation safety practices.

ELIGIBILITY:
Inclusion Criteria:

* active members of American Academy of Pediatric Dentistry

Exclusion Criteria:

* pre and post doctoral students and affiliated members

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6473 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Behavioral Change | Day 1
  The primary outcome of this study is the change in pediatric dentists' reported willingness to adopt rectangular collimation based on the nudging strategies employed. Specifically, the study will measure whether pictorial framing and traffic-light-color-coding influence the likelihood of adopting rectangular collimation in clinical practice. Responses collected in 10 point visual analog scale will be compared for effectiveness of each nudging strategy individually in promoting behavior change and mean scores will be compared across all groups.

CONTACTS AND LOCATIONS:
Overall Officials: Hashim Nainar, Dentist, Study Director — University of Toronto
Locations (1):
- Faculty of Dentistry, University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
It does not abide by the requirements laid out by American Academy of Pedaitric Dentistry, which provided the participant list. Individual partipants are not consenting to sharing of individual data.

REFERENCES:
- [Background] Oakes AH, Patel MS. A nudge towards increased experimentation to more rapidly improve healthcare. BMJ Qual Saf. 2020 Mar;29(3):179-181. doi: 10.1136/bmjqs-2019-009948. Epub 2019 Nov 19. No abstract available. PMID 31744847
- [Background] Schubbe D, Scalia P, Yen RW, Saunders CH, Cohen S, Elwyn G, van den Muijsenbergh M, Durand MA. Using pictures to convey health information: A systematic review and meta-analysis of the effects on patient and consumer health behaviors and outcomes. Patient Educ Couns. 2020 Oct;103(10):1935-1960. doi: 10.1016/j.pec.2020.04.010. Epub 2020 May 11. PMID 32466864